CLINICAL TRIAL: NCT02215226
Title: Establishing a Sero-correlate of Protection Against Invasive Group B Streptococcus Disease in Newborns and Young Infants Aged <=90 Days
Brief Title: GBS Sero-correlate of Protection
Acronym: V98_28OBTP
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Principal Investigator, Shabir Madhi, Medical officer, University of Witwatersrand, South Africa
Other Study IDs: V98_28OBTP
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Invasive Group B Streptococcus Disease
Keywords: Group B Streptococcus, early onset disease, late onset disease, anticapsular antibodies, serotype specific
MeSH Terms: conditions — Late Onset Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Cord blood and maternal blood (serum samples) Vaginal swab samples from mothers Invasive GBS isolates from cases
Oversight: Data Monitoring Committee: No

SUMMARY:
Compare anticapsular antibody levels against Group B Streptococcus at delivery in mothers and their infants who develop disease versus those who do not. Use this comparison to establish antibody levels associated with reductions in risk of GBS disease in infants aged less than 90 days.

DETAILED DESCRIPTION:
Group B Streptococcus (GBS) is a leading cause of invasive disease during the neonatal period in developed and developing countries. The global incidence of disease is 0.53 per 1000 live births, though a substantially higher incidence has been reported from South Africa (3 per 1000 live births). Of the disease-causing serotypes, types Ia and III account for over 70% of invasive disease in young infants. The introduction of screening for maternal rectovaginal GBS colonization, with subsequent treatment of colonized women with intrapartum antibiotic prophylaxis (IAP) at delivery, has led to a >80% reduction in the incidence of disease in some settings (Schrag, 2012). However, the residual burden of early-onset disease (EOD) in countries which have implemented universal screening and IAP remains similar to the incidence of late-onset disease (LOD), which has not declined over time. The resources necessary to implement a screening and IAP program has limited the establishment of this intervention in other developed and most developing countries.

GBS capsular polysaccharide-protein conjugate vaccines (GBS-CV) aimed at the immunization of pregnant women, with protection of the newborn expected from trans-placental acquisition of the induced antibodies in utero have been developed.

There are a number of challenges to undertaking a large efficacy trial of GBS-CV aimed at licensure of this vaccine. Consequently, licensure of GBS-CV may depend on establishing an immunologic/serologic correlate of protection against invasive disease in newborns, as has been successfully motivated for and adopted in the licensure pathway of meningococcal vaccines. Although previous studies have aimed to identify serotype-specific correlates of anticapsular antibody protection against invasive GBS disease during early-infancy; differences in study-design, age-range of invasive-cases, antibody assay methods and a lack of standardized reference serum between tests mean a robust sero-correlate of protection against GBS has yet to be identified.

We propose to conduct a case control study nested within a prospective, longitudinal cohort of mothers and their infants <=90 days of age, at one academic hospital center in South Africa. The limited intrapartum antibiotic exposure (10-12% deliveries), relatively high incidence of both EOD and LOD (2 per 1000 live births and 1 per 1000 live births respectively) and standardized laboratory surveillance (for case identification) offers an optimal setting in which to establish correlates of protection against the GBS serotypes that predominate in this setting (serotypes Ia and III for EOD and serotype III for LOD).

ELIGIBILITY:
Inclusion Criteria:

* (i) Pregnant women attending participating community/hospital antenatal clinics and/or delivering at participating delivery centers.

(ii) Subjects aged ≥18 years. (iii) Able to understand and comply with planned study procedures. (iv) Provides written informed consent.

Exclusion Criteria:

* (i) Refuses to consent to study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women aged 18 years or older attending for antenatal care or delivery at Chris Hani Baragwanath Academic hospital, and infants who develop GBS disease at the other 2 hospitals in the Johannesburg area
Sampling Method: Non-Probability Sample
Enrollment: 35274 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Risk of early onset Group B Steptococcus disease (due to serotypes Ia or III) with respect to maternal or newborn anticapsular antibody levels at delivery. | Birth to 6 days of age
  Early onset Group B Streptococcus disease due to serotypes Ia & III

SECONDARY OUTCOMES:
Risk of late onset Group B Streptococcus disease (due to serotypes III) with respect to maternal or newborn anticapsular antibody levels at delivery | 7 to 90 days
  Late onset Group B Streptococcus disease due to serotype III

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory and Meningeal Pathogen Research Unit, Soweto, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Derived] Gent V, Dhar N, Izu A, Jones S, Dangor Z, Briner C, Hosken N, Kwatra G, Madhi SA. Association of serum anti-gbs2106 protein immunoglobulin G (IgG) in newborns and risk reduction of invasive group B streptococcus disease during early infancy. Vaccine. 2025 Apr 30;54:127016. doi: 10.1016/j.vaccine.2025.127016. Epub 2025 Mar 14. PMID 40088514
- [Derived] Madhi SA, Izu A, Kwatra G, Jones S, Dangor Z, Wadula J, Moultrie A, Adam Y, Pu W, Henry O, Briner C, Cutland CL. Association of Group B Streptococcus (GBS) Serum Serotype-Specific Anticapsular Immunoglobulin G Concentration and Risk Reduction for Invasive GBS Disease in South African Infants: An Observational Birth-Cohort, Matched Case-Control Study. Clin Infect Dis. 2021 Sep 7;73(5):e1170-e1180. doi: 10.1093/cid/ciaa1873. PMID 33341870
- [Derived] Jallow S, Agosti Y, Kgagudi P, Vandecar M, Cutland CL, Simoes EAF, Nunes MC, Suchard MS, Madhi SA. Impaired Transplacental Transfer of Respiratory Syncytial Virus-neutralizing Antibodies in Human Immunodeficiency Virus-infected Versus -uninfected Pregnant Women. Clin Infect Dis. 2019 Jun 18;69(1):151-154. doi: 10.1093/cid/ciy1071. PMID 30561563